CLINICAL TRIAL: NCT07161869
Title: Preoperative Evaluation of Lymph Nodes of Cholangiocarcinoma by Endoscopic Ultrasound (POELH-III)
Brief Title: Preoperative Evaluation of Lymph Nodes of Cholangiocarcinoma (POELH-III)
Acronym: POELH-III
Status: Not yet recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Lydi M.J.W. van Driel, MD, MSc, PhD, Principal Investigator, Erasmus Medical Center
Other Study IDs: MEC-2022-0402.1
Record Dates: First submitted 2025-08-28; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Hilar Cholangiocarcinoma; Intrahepatic Cholangiocarcinoma (Icc); Cholangiocarcinoma; Perihilar Cholangiocarcinoma; Common Bile Duct Neoplasms; Adenocarcinoma of Biliary Tract
Keywords: poelh; EUS; Lymph node; cholangiocarcinoma; biliary tract cancer
MeSH Terms: conditions — Klatskin Tumor; Cholangiocarcinoma; Cirrhosis, Familial, with Pulmonary Hypertension; Common Bile Duct Neoplasms; Biliary Tract Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Presumed resectable perihilar, intrahepatic or mid-common bile duct (CBD) cholangiocarcinoma
  Interventions: Procedure: Registration of all findings during preoperative Endoscopic Ultrasound

INTERVENTIONS:
Procedure: Registration of all findings during preoperative Endoscopic Ultrasound — Using the improved POELH-III EUS format

SUMMARY:
In the POELH-II trial (Clinicaltrials.gov ID NCT05678218) patients with presumed resectable perihilar (pCCA), intrahepatic (iCCA) or mid-common bile duct (CBD) cholangiocarcinoma had the outcomes of their preoperative endoscopic ultrasound (EUS) registered. This EUS procedure was done systematically, targeting lymph nodes (LNs) with the aim to identify LN metastases preoperatively.

The goal of this follow-up observational cohort study (POELH-III) is to assess the yield of preoperative EUS, with an improved EUS approach. The EUS protocol as used in the POELH-II trial was improved based on preliminary results of the POELH-II trial. The main questions it aims to answer is:

- The number of patients precluded from surgical work-up due to positive regional or extraregional LNs identified by EUS guided tissue acquisition

ELIGIBILITY:
Inclusion Criteria:

* Presumed resectable pCCA OR
* Presumed resectable iCCA OR
* Presumed resectable mid-common bile duct CCA OR
* Presumed unresectable pCCA worked-up for Liver Transplantation AND
* Written informed consent must be given according to International Council on Harmonisation/Good Clinical Practice guidelines, and national/local regulations AND
* Age > 18 years.

Exclusion Criteria:

* Patients with a history of treated CCA
* Patients with CCA for which a pancreatoduodenectomy is indicated, based on cross-sectional imaging
* Patients with a history of treated liver malignancy
* Patients with a contra-indication for EUS-tissue acquisition (f.e. uncorrectable coagulopathy or platelet disorder), in line with current clinical practice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected iCCA or pCCA who have a presumed resectable carcinoma will be invited to participate. Patients with CCA distal from the cystic junction but proximal from the pancreatic body are eligible for inclusions as well, as treatment is similar to Bismuth I pCCA. In other words, all patients with CCA that is not distal CCA for which a pancreato-duodenectomy is indicated, are eligible for inclusion. Also patients with presumed unresectable pCCA who are worked-up for liver transplantation are invited to participate. At time of inclusion a definitive diagnosis of iCCA/pCCA is not obligatory, since definitive diagnosis of CCA is sometimes confirmed during the preoperative EUS through EUS guided biopsy of the mass. The probable diagnosis of iCCA/pCCA and the suspected resectability will be established during the multidisciplinary meeting, based on clinical symptoms, cross-sectional imaging, endoscopy and laboratory tests.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
The number of patients precluded from surgical work-up due to positive regional or extraregional lymph nodes identified by endoscopic ultrasound guided tissue acquisition | Through study completion, max 1 year

SECONDARY OUTCOMES:
Short term and long term complications of the EUS (+/- tissue acquisition) procedure | Through study completion, max 1 year
  Short term (<30 days)
  * Sedation related: consisting of cardiovascular-related complications (cardiac arrhythmias, myocardial ischemia/infarction), respiratory- related complications (respiratory depression, hypoxia, airway obstruction, pulmonary aspiration of gastric contents) and allergic reactions.
  * Hemorrhage (outside peritoneal wall): defined as clinical evidence of bleeding with a hemoglobin drop of >3g/dl with the need for resuscitation or additional intervention
  * Perforation: defined as evidence of air or luminal contents outside the gastro-intestinal tract together with clinical symptoms, requiring percutaneous drainage or surgery
  * Mortality
  Long term (>30 days)
  - Tumor seeding; defined as proof of carcinoma in the biopsy tract during follow-up or at autopsy

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC University Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Background] Larghi A, Rimbas M, Ardito F, Rizzatti G, Giuliante F. Letter to the Editor: EUS-FNA for Lymph Nodes Staging in Cholangiocarcinoma: Should It Become Standard of Care? Hepatology. 2020 Oct;72(4):1496. doi: 10.1002/hep.31266. No abstract available. PMID 32277489
- [Background] Malikowski T, Levy MJ, Gleeson FC, Storm AC, Vargas EJ, Topazian MD, Abu Dayyeh BK, Iyer PG, Rajan E, Gores GJ, Roberts LR, Chandrasekhara V. Endoscopic Ultrasound/Fine Needle Aspiration Is Effective for Lymph Node Staging in Patients With Cholangiocarcinoma. Hepatology. 2020 Sep;72(3):940-948. doi: 10.1002/hep.31077. Epub 2020 Jul 9. PMID 31860935
- [Background] Gleeson FC, Rajan E, Levy MJ, Clain JE, Topazian MD, Harewood GC, Papachristou GI, Takahashi N, Rosen CB, Gores GJ. EUS-guided FNA of regional lymph nodes in patients with unresectable hilar cholangiocarcinoma. Gastrointest Endosc. 2008 Mar;67(3):438-43. doi: 10.1016/j.gie.2007.07.018. Epub 2007 Dec 3. PMID 18061597
- [Background] de Jong DM, van de Vondervoort S, Dwarkasing RS, Thomeer MGJ, Doukas M, Voermans RP, Verdonk RC, Polak WG, de Jonge J, Bruno MJ, Van Driel LMJW, Groot Koerkamp B. Endoscopic ultrasound with tissue acquisition of lymph nodes in patients with potentially resectable intrahepatic cholangiocarcinoma. Endosc Int Open. 2024 Aug 23;12(8):E998-E1005. doi: 10.1055/a-2366-2592. eCollection 2024 Aug. PMID 39184062
- [Background] de Jong DM, den Hoed CM, Willemssen FEJA, Thomeer MGJ, Bruno MJ, Koerkamp BG, de Jonge J, Alwayn IPJ, van Hooft JE, Hoogwater F, van der Heide F, Inderson A, van Vilsteren FGI, van Driel LMJW. Impact of EUS in liver transplantation workup for patients with unresectable perihilar cholangiocarcinoma. Gastrointest Endosc. 2024 Apr;99(4):548-556. doi: 10.1016/j.gie.2023.10.047. Epub 2023 Oct 27. PMID 37890597
- [Background] de Jong DM, van de Vondervoort S, Dwarkasing RS, Doukas M, Voermans RP, Verdonk RC, Polak WG, de Jonge J, Koerkamp BG, Bruno MJ, van Driel LMJW. Endoscopic ultrasound in patients with resectable perihilar cholangiocarcinoma: impact on clinical decision-making. Endosc Int Open. 2023 Feb 2;11(2):E162-E168. doi: 10.1055/a-2005-3679. eCollection 2023 Feb. PMID 36741342
- [Background] de Jong DM, Lammers WJ, van Driel LMJW. Time to standardize preoperative EUS for lymph node staging in resectable extrahepatic cholangiocarcinoma. J Hepatol. 2025 Dec;83(6):e290-e291. doi: 10.1016/j.jhep.2025.06.031. Epub 2025 Jul 9. No abstract available. PMID 40645595